CLINICAL TRIAL: NCT06237842
Title: Evaluation of Wearable Technologies for Sleep Monitoring in Children and Adolescents
Brief Title: Wearable Technologies for Sleep in Children and Adolescents
Status: Recruiting | Type: Observational
Sponsor: SleepUp Tecnologia em Saúde Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: SleepUp_#03
Record Dates: First submitted 2024-01-23; First posted 2024-02-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sleep; Pediatric Sleep Apnea
Keywords: Pediatric sleep; Adolescent sleep; EEG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy participants: Participants from 3 to 18 years old, from both genders and with no sleep disorders
  Interventions: Diagnostic Test: Diagnostic Test: EEG headband+Ring oximeter (RO)+Actigraphy (ACT)
- Participants with sleep disorders: Participantes with one sleep disorder or complaint.
  Interventions: Diagnostic Test: Diagnostic Test: EEG headband+Ring oximeter (RO)+Actigraphy (ACT)

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: EEG headband+Ring oximeter (RO)+Actigraphy (ACT) — Combination of ACT+RO+EEG. This is not an intervention, but rather a combination of devices to be tested regarding its diagnostic validity.

SUMMARY:
This study aims to evaluate the viability of wearable and portable technologies for sleep staging in children and adolescents. The results will be compared with polysomnography, in order to achieve clinical and diagnostic validation. Three domains of devices will be used: movement sensors, wearable EEG band and pulse oximetry.

The project will include individuals between the ages of 3 and 18 who reside in São Paulo city and undergo a polysomnography test at the Sleep Laboratory of the Children's Institute of the Hospital das Clínicas of the University of São Paulo.

DETAILED DESCRIPTION:
This study aims to evaluate the viability of the combined use of wearable and portable technologies for sleep staging. The results will be compared with polysomnography, in order to achieve clinical and diagnostic validation. Three domains of devices will be used:

* Movement sensors: Devices equipped with movement sensors (such as an accelerometer) able to monitor movement over the using period, converting this information in data related to the sleep-wakefulness cycle. In this category, the reference devices are the actimeters/actigraphs (ACT). Its use is recommended by the American Academy of Sleep Medicine to the diagnosis of insomnia and circadian sleep disorders, and should be used for 3 to 14 consecutive days. Other wearable devices, such as smartwatches, are also used with the same purpose, although not validated for clinical use.
* Wearable EEG band: EEG is a mandatory feature for type-1 polysomnography and a requirement for regular sleep staging. The project will utilize a wearable EEG band in combination with actigraphy and a ring oximeter to improve the estimation of sleep stages. This study will test wearable EEG bands with the following minimal specifications: dry EEG electrodes (no need for paste, gel, or other conductors), presented as a headband or stripe, a minimal sampling rate of 500Hz, noise, high and low filters, a battery lasting at least 8 hours, a maximum weight of 200g (including the whole device), and support for Bluetooth connection.
* Ring oximeter: The project will utilize a ring oximter to record the overnight blood oxygen levels, heart rates, and body movements.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* 3 to 18 years olnde
* Resident in the city of São Paulo
* Candidate to perfome a polysomnography test at the Sleep Laboratory of the Children's Institute of the Hospital das Clínicas of the University of São Paulo.

Exclusion Criteria:

* None.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children/adolescents who come to the Sleep Laboratory of the Children's Institute of the University of São Paulo for a polysomnography test.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Latency | Immediately after the polysomnography.
  Time from the beginning of the polysomnographic record until the first epoch of sleep.
Total sleep time | Immediately after the polysomnography.
  Total time of epochs staged as sleep.
Sleep efficiency | Immediately after the polysomnography.
  Percentage of sleep in relation to total record/bed time.
Wake after sleep onset | Immediately after the polysomnography.
  Total time of epochs staged as "wake" after sleep latency.
Latency to REM sleep | Immediately after the polysomnography.
  Time from sleep latency until the first epoch of REM sleep.
Total time for each sleep stage | Immediately after the polysomnography.
  Time corresponding to epochs staged as each of the sleep stages (N1, N2, N3 and REM)
Percentage each sleep stage | Immediately after the polysomnography.
  Percentage corresponding to epochs staged as each of the sleep stages (N1, N2, N3 and REM), in comparison with total sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Soster, PhD, Principal Investigator — Instituto da Criança do Hospital da Clínicas- FMUSP; Anna Monazzi, PhD, Study Director — Instituto da Criança do Hospital da Clínicas- FMUSP
Locations (1):
- Instituto da Criança do Hospital da Clínicas - FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The dissemination of Individual Participant Data (IPD) from this study is strictly limited by restrictions on the release of intellectual property, concerns regarding participant privacy and confidentiality, and the absence of explicit consent for extensive data sharing. However, upon reasonable request and subject to approval by the study's principal investigator, anonymized datasets may be provided to qualified researchers. It is imperative that requests include a thorough research proposal and a rationale that substantiates the need for the resources in question.